CLINICAL TRIAL: NCT05461768
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, and Preliminary Efficacy of BL-M07D1injection in Patients With Locally Advanced or Metastatic HER2-positive/Low-expression Breast Cancer and Other Solid Tumors
Brief Title: A Study of BL-M07D1 in Patients With Locally Advanced or Metastatic HER2 Positive/Low Expression Breast Cancer and Other Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: SystImmune Inc. (Industry); Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-M07D1-101
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Locally Advanced or Metastatic Solid Tumor
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive BL-M07D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M07D1

INTERVENTIONS:
Drug: BL-M07D1 — Administration by intravenous infusion

SUMMARY:
In phase Ia study, the safety and tolerability of BL-B07D1 in patients with locally advanced or metastatic HER2-positive/low-expression breast cancer and other solid tumors will be investigated to determine the dose-limiting toxicity (DLT), maximum tolerated dose (MTD) of BL-M07D1.

In phase Ib study, the safety and tolerability of BL-M07D1 at the phase Ia recommended dose will be further investigated, and recommended phase II dose (RP2D) for phase II clinical studies will be determined.

In addition, the preliminary efficacy, pharmacokinetic characteristics, and immunogenicity of BL-M07D1 in patients

ELIGIBILITY:
Inclusion Criteria:

* 1. Sign the informed consent voluntarily and follow the program requirements
* 2. No gender limitation;
* 3. Age: ≥18 years old and ≤75 years old (Stage Ia);≥18 years old (Ib);
* 4. Expected survival time ≥3 months;
* 5. Inoperable locally advanced or metastatic HER2-positive/low-expression breast cancer and other solid tumors that have been histopathologically and/or cytologically confirmed and have failed standard therapy, or are not available for standard therapy, or are not currently eligible for standard therapy; HER2 positive: IHC3+, or IHC2+ and ISH positive; HER2 low expression: IHC2+ and ISH negative, or IHC1+;
* 6. Agree to provide archived tumor tissue samples or fresh tissue samples from the primary tumor or metastatic tumor within 2 years (to detect the expression of HER2 protein in tumor pathological tissue and explore the correlation between HER2 protein and bl-M07D1 validity index); If subjects are unable to provide tumor tissue samples, they will be admitted after evaluation by the investigator if other admission criteria are met.
* 7. Must have at least one measurable lesion as defined by RECIST V1.1;
* 8. ECOG score of 0 or 1;
* 9. Toxicity of previous antitumor therapy has returned to level ≤1 as defined by NCI-CTCAE V5.0 (the investigator considered asymptomatic laboratory abnormalities, such as elevated ALP, hyperuricemia, and elevated blood glucose, etc.); Except for toxicity that the investigator judged to have no safety risk, such as alopecia, pigmentation, grade 2 peripheral neurotoxicity, etc.);
* 10. No serious cardiac dysfunction, left ventricular ejection fraction ≥50%;
* 11. Organ function level must meet the following requirements and meet the following standards: A) Bone marrow function: absolute neutrophil count (ANC) ≥1.5×10^9/L, platelet count ≥90×10^9/L, hemoglobin ≥90 g/L; B) Liver function: total bilirubin (TBIL≤1.5 ULN), AST and ALT ≤2.5 ULN in patients without liver metastasis, AST and ALT ≤5.0 ULN in patients with liver metastasis; C) Renal function: creatinine (Cr) ≤1.5 ULN, or creatinine clearance (Ccr) ≥50 mL/min (according to the Cockcroft and Gault formula).
* 12. Coagulation function: International standardized ratio (INR) ≤1.5, and activated partial thrombin time (APTT) ≤1.5ULN;
* 13. Urinary protein ≤2+ or ≤1000mg/24h;
* 14. For premenopausal women at risk of fertility, pregnancy tests must be performed within 7 days prior to the start of treatment. Serum/urine pregnancy must be negative and must be non-lactation; All enrolled patients (male and female) should use adequate barrier contraception throughout the treatment cycle and 6 months after the end of treatment

Exclusion Criteria:

* 1. Prior use of chemotherapy, biotherapy, immunotherapy, radical radiotherapy, major surgery (as defined by the investigator), targeted therapy (including small molecule tyrosine kinase inhibitors) and other antitumor therapies within 4 weeks or 5 half-lives (whichever is less) prior to initial dosing; Mitomycin and nitrosourea were administered within 6 weeks prior to initial administration; For oral fluorouracil drugs such as gio, capecitabine, or palliative radiotherapy within 2 weeks before initial administration; The Chinese medicine with anti-tumor indication was given within 2 weeks before the first administration.
* 2. Prior ADC treatment (phase Ib only) with the toxin of camptothecin derivatives (topoisomerase I inhibitors);
* 3. History of severe heart disease, such as symptomatic congestive heart failure (CHF) grade 2 or greater (CTCAE 5.0), NYHA grade 2 or greater heart failure, history of transmural myocardial infarction, unstable angina, etc.;
* 4. QT prolongation (male QTc > 450 msec or female QTc > 470 msec), complete left bundle branch block, III atrioventricular block;
* 5. Active autoimmune diseases and inflammatory diseases, such as: systemic lupus erythematosus, systemic treatment of psoriasis, rheumatoid arthritis, inflammatory bowel disease, and hashimoto's thyroiditis, etc., with the exception of type I diabetes, only replacement therapy can control the hypothyroidism, no systemic treatment of skin disease (e.g., vitiligo, psoriasis);
* 6. Other malignancies diagnosed within 5 years prior to first administration, except for radical basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or radical resected carcinoma in situ;
* 7. Screening for unstable thrombotic events such as deep vein thrombosis, arterial thrombosis and pulmonary embolism requiring therapeutic intervention within the first 6 months; Infusion device-related thrombosis is excluded;
* 8. Patients with poorly controlled pleural effusion with clinical symptoms were judged by researchers to be unsuitable for inclusion;
* 9. Hypertension poorly controlled by medications (systolic & GT; 150 mmHg or diastolic pressure & GT; 100 mmHg);
* 10. According to CTCAE V5.0, patients were defined as ≥3 grade of lung disease, ≥2 grade of radioactive lung disease, existing or with a history of ILD;
* 11. Symptoms of active CNS metastasis. But the researchers concluded that patients with stable parenchymal metastases could be included. The definition of stability must meet the following four requirements: A. Seizureless state lasting > 12 weeks with or without antiepileptic drugs; B. Glucocorticoids are not required; C. Two consecutive MRI scans (at least 4 weeks between scans) showed stable imaging state; D. Asymptomatic patients have been stable for more than 1 month after treatment;
* 12. Patients with a history of allergy to recombinant humanized antibody or human-mouse chimeric antibody or to any excipient component of BL-M07D1;
* 13. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation (ALLO-HSCT);
* 14. Equivalent cumulative dose of doxorubicin in anthracycline adjuvant therapy was > 360 mg/m^2;
* 15. Positive human immunodeficiency virus antibody (HIVAb), active tuberculosis, active hepatitis B virus infection (HBV-DNA copy number > lower limit) or active hepatitis C virus infection (HCV antibody positive and HCV-RNA > lower limit);
* 16. Active infections requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis, etc.
* 17. Participated in another clinical trial within 4 weeks prior to initial administration (starting from the time of last administration);
* 18. Pregnant or nursing women;
* 19. Other conditions considered inappropriate for participation in this clinical trial by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-08-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose limiting toxicity (DLT) | Up to 21 days after the first dose
  The DLT observation period was the first treatment period for each dose level, and the DLT observation period was extended if there was a delay in administration .
Phase Ia: Maximum tolerated dose (MTD) | Up to 21 days after the first dose
  In the dose escalation stage, MTD was selected as the highest dose whose DLT rate estimate was closest to the target DLT rate, but did not exceed the upper bound of the EQUIVALENT interval of DLT rate.
Phase Ib: Phase II clinical study recommended dose (RP2D) | Up to 21 days after the first dose
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-M07D1

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B07D1 . The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M07D1 .
Cmax | Up to 21 days after the first dose
  Maximum serum concentration (Cmax) of BL-M07D1 will be investigated
T1/2 | Up to 21 days after the first dose
  Half-life (T1/2) of BL-M07D1 will be investigated.
AUC0-t | Up to 21 days after the first dose
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration
Tmax | Up to 21 days after the first dose
  Time to maximum serum concentration (Tmax) of BL-M07D1 will be investigated
CL (Clearance) | Up to 21 days after the first dose
  CL in the serum of BL-M07D1 per unit of time will be investigated.
Ctrough | Up to 21 days after the first dose
  Ctough is defined as the lowest serum concentration of BL-M07D1 prior to the next dose will be administered.
ADA (anti-drug antibody) | Up to approximately 24 months
  Incidence and titer of ADA of BL-M07D1 will be evaluated.
Nab (neutralizing antibody) | Up to approximately 24 months
  Incidence and titer of Nab of BL-M07D1 will be evaluated
Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of Response (DOR) Duration of Response (DOR) Duration of Response (DOR) Duration of Response (DOR) Duration of Response (DOR) Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Progression-free Survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of BL-B07D1 to the first date of either disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Erwei Song, PHD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Herui Yao, PHD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (7):
- China (7):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangdong, Guangzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Jinan Central Hospital, Jinan, Shandong
  - Run Run Shaw Hospital Affiliated to Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No